CLINICAL TRIAL: NCT04023968
Title: Effects of Two Psychosocial Wellness Workshops on Sleep, Stress Management and Well-being: Exploration of Psychophysiological Mechanisms
Brief Title: Student Wellness Workshop Study
Acronym: SWW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1508074542A003
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Stress; Stress, Psychological; Stress Reaction; Adjustment; Adjustment, Social; Adjustment, Emotional
MeSH Terms: conditions — Stress, Psychological; Fractures, Stress; Social Adjustment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YESplus workshop (Experimental): Your Enlightened Side, plus more (YESplus) is an four-day, 15-hour integrative life skills workshop with a strong emphasis on breathing techniques and social connectedness. In addition to specific contemplative techniques such as yoga, mindfulness meditation, and compassion meditation that help cultivate inner peace, YESplus incorporates discussions and other activities to facilitate social connectedness, leadership, and community service. During the workshop, participants have ample time to learn and practice the Sudarshan Kriya Yoga (SKY) technique, as well as to ask questions. SKY has four sequential, form- and rhythm-specific breathing components interspersed with normal breathing while sitting in a relaxed position with eyes closed, followed by Yoga Nidra. A certified instructor with a minimum of 1,000 hours of SKY instruction training will lead each workshop.
  Interventions: Behavioral: YESplus workshop
- WOW! workshop (Active Comparator): A comparison workshop titled "Wisdom On Wellness" (WOW!) will be implemented to control for potential expectancy effects, time commitment, group-based interactions, and wisdom/knowledge of YESplus that is anticipated to have beneficial effects on stress management and well-being, allowing for more rigorous evaluation of the contemplative practices and other activities unique to the YESplus workshop. This workshop differs from YESplus due to the increased focus on cognitive approaches to conceptualizing and managing stress (e.g. thoughts about the past and future versus present moment), and absence of physical or somatic activities.
  Interventions: Behavioral: WOW! workshop

INTERVENTIONS:
Behavioral: YESplus workshop — See description in "Arms" section.
  Arms: YESplus workshop
Behavioral: WOW! workshop — See description in "Arms" section.
  Arms: WOW! workshop

SUMMARY:
While efficacy of Sudarshan Kriya Yoga (SKY) has been demonstrated in a number of prior studies, little is known about the effects of SKY taught as part of the Your Enlightened Side (YESplus) workshop designed for college students. Thus, this study aims to assess the effects of YESplus on well-being, including sleep patterns, and physiological stress response.

DETAILED DESCRIPTION:
The transition from adolescence to adulthood, particularly for college students, is accompanied by several major life changes and challenges. For many individuals, this is a period when one moves away from home, begins interacting with different peer groups, and has greater financial and academic responsibilities. The emotional stress associated with these changes is correlated with less time devoted to sleep, increased alcohol intake reduced academic performance and increased rates of anxiety disorders and/or depression.

Your Enlightened Side (plus more) (YESplus) is a life skills workshop with a strong emphasis on breathing practices for reducing stress and increasing well-being. Additional stress management tools including meditation, yoga, and interpersonal exercises that impart social emotional learning skills and stress reduction strategies complement the breathing techniques.

The central practice taught in YESplus is a unique rhythmical breathing technique called Sudarshan Kriya. It is taught along with two preparatory breathing practices: an advanced form of Ujjayi breathing (breathing against airway resistance) and bhastrika (forceful nasal breathing). Collectively, these three breathing practices are referred to as Sudarshan Kriya Yoga (SKY).

Prior literature has demonstrated significant improvements in psychological and physiological outcomes of SKY in adults, including decreases in subjective stress, clinical and subclinical depression and anxiety, posttraumatic stress symptoms,impulsivity, and tobacco use, as well as increases in calm, mental focus, emotion regulation, and overall well-being.

However, little is known about the effects of SKY specifically taught in the YESplus workshop format designed for college students. One randomized controlled trial has demonstrated attenuated levels of subjective stress and several hematological parameters, including lymphocytes and platelet count, during exam periods following SKY training. These findings have not yet been replicated, and the extent to which the effects of YESplus generalize to other health-related changes such as cardiovascular function remain unclear.

Addressing the gap in the literature described above and to provide further preliminary data on the specific effects of YESplus on well-being and stress physiology, this study aims to evaluate measures of self-reported wellness across a variety of questionnaires, in addition to changes in heart rate variability and salivary cortisol levels with a stress induction task. To control for expectancy effects, overall time spent with the workshop, social contact, and exposure to cognitive stress management strategies that may influence the observed effects of YESplus not specific to the yogic breathing and deep social connectedness at the core of the YESplus targets, a comparison workshop with all of these potential supplementary contributors will be included, titled "Wisdom On Wellness" (WOW!).

Participation will include three laboratory visits at pre-workshop (T1), post-workshop (T2), and 1-2 month follow-up (T3) time points and four workshop sessions described below.

Screening: Interested participants will first be directed to an online pre-screening survey. The survey will begin with a prompt describing the study and requiring understanding via checkbox that the survey is for screening purposes. The survey will collect information such as name, e-mail address, date of birth, motivation for the study, student status, prior contemplative practice experience, ability to meet the time commitment, panic and bipolar symptoms, and potential affiliation with other participants. If any of the exclusion criteria indicated above are met, the participant will be notified of ineligibility.

Enrollment and randomization: Eligible participants will be first grouped in clusters with any other participants with known affiliations stated in the online screener, in order to minimize possibility of learning about material of the other workshop, then assigned a workshop via random number generator.

Laboratory Visits: In-person laboratory visits will be conducted at the University of Arizona Respiratory Physiology Laboratory on the main UA campus. Workshops will be conducted in various buildings on the main UA campus depending on reservation availability.

Actigraphy, sleep diary, online questionnaires and practice logs measures will be completely remotely after the instruments are provided to participants during an in-laboratory visit.

In addition to actigraphy, sleep diary, online questionnaires, and home practice logs (for T2 and T3 time points) the following data will be collected during each laboratory visit: electrocardiography (ECG) with concurrent respiratory inductance plethysmography (RIP) and pulse oximetry recordings, as well as salivary cortisol at baseline, post-stress induction task, 30-min post-stress-induction-onset, and 45-min post. ECG, RIP belts, and pulse oximetry will be recorded continuously, in addition to the designated resting recording periods.

Workshop evaluations: Both workshop participants and instructors will complete a brief questionnaire at two time points (end of Day 1 and end of Day 4) during the workshop to indicate expectation of workshop benefit.

Stress Induction. The Maastricht Acute Stress Test (MAST), a previously described and increasingly used stress induction task will be utilized. A research staff member in a white laboratory coat will explain that the session will be video-recorded to then be coded afterwards by trained raters, provide background information regarding performance norms, and express an expected ability of the participant to perform comparably. Next, the researcher will provide instructions for the task that will be guided by a Powerpoint presentation. The MAST consists of a 10 minute acute stress phase that combines elements of both the commonly used Cold Pressor Test and Trier Social Stress Test, adding an element of uncertainty by cycling between these two tests at slightly unpredictable time intervals. For the hand immersion trials (HIT), participants will insert their dominant hand and wrist in a bucket of ice water (approximately 2° C) for up to 90 seconds. Participants are instructed they may remove their hand at any time. Upon removal, participants will place their hand on a towel and immediately begin a serial subtraction task, for which participants will be instructed to count backwards by 13, 17, or 18 from a randomly selected number between 2013 and 2073, with interjections to start over from the beginning if any calculations are incorrect. Neutral or negative feedback will be provided throughout the task, including comments such as "That's wrong. Start over" and "You're going too slowly."

ELIGIBILITY:
Inclusion Criteria:

* Current identification with student status, which may include undergraduate, graduate, continuing studies, or post-baccalaureate/pre-doctoral.

Exclusion Criteria:

* No history of panic disorder, psychosis, or mania (with or without psychotic features), which may be risk factors for adverse effects of the yogic breathing intervention. These symptoms will be pre-screened via online questionnaire. The use of psychoactive medication will be monitored via sleep diary.
* No current substance dependence, assessed via online self-report pre-screening questionnaire.
* No current use of medications with known effects on sleep or stress physiology including antidepressants (SSRI, SNSI, NDRI, atypical, TCA, MAOI), anitpsychotics, benzodiazepines, non-benzodiazepine receptor agonists, melatonin and melatonin receptor agonists, orexin/hypocretin receptor antagonists, barbiturates, mood stabilizers, anticonvulsants, anticholinergics, first generation antihistamines, and stimulants including NRI, antihypertensives, opioids, or systemic (non-topical) corticosteroids.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS) from baseline to post-intervention | 3 months
  self-report questionnaire; range: 0-40, higher scores indicate higher perceived stress
Change in Pittsburgh Sleep Quality Index (PSQI) from baseline to post-intervention | 3 months
  self-report questionnaire; range: 0-21, higher scores indicate higher sleep disturbance
Change in Social Connectedness (SC) from baseline to post-intervention | 3 months
  self-report questionnaire; range: 20-120, higher scores indicate higher perceived social connectedness
Change in Resting heart rate variability (HRV) from baseline to post-intervention | 3 months
  2 min average HRV at beginning of each laboratory visit
Change in HRV reactivity to stress induction from baseline to post-intervention | 3 months
  average HRV during stress induction, minus baseline from that laboratory visit
Change in HRV recovery from stress induction from baseline to post-intervention | 3 months
  average HRV 30 min after stress induction, minus baseline from that laboratory visit

SECONDARY OUTCOMES:
Change in Mood and Anxiety Symptom Questionnaire (MASQ) from baseline to post-intervention | 3 months
  self-report questionnaire; range: 26-130, higher scores indicate higher severity of mood symptoms
Change in Big Five personality inventory (BFI) subscale scores from baseline to post-intervention | 3 months
  self-report questionnaire; subscales include the following, with higher scores indicating higher levels of the descriptive name: Extraversion (range: 8-40), Agreeableness (range: 9-45); Conscientiousness (range: 9-45); Neuroticism (range: 8-40); Openness (range: 10-50);
Change in Rosenberg Self-Esteem Scale (RSES) from baseline to post-intervention | 3 months
  self-report questionnaire; range: 0-30, higher scores indicate higher self-esteem
Change in Satisfaction With Life Scale (SWL) from baseline to post-intervention | 3 months
  self-report questionnaire; range: 5-35, higher scores indicate higher satisfaction with life
Change in Heart Rate (HR) from baseline to post-intervention | 3 months
  following same analysis approach as HRV
Change in Respiratory Rate (RR) from baseline to post-intervention | 3 months
  following same analysis approach as HRV
Change in Respiratory Sinus Arrhythmia (RSA) from baseline to post-intervention | 3 months
  following same analysis approach as HRV

CONTACTS AND LOCATIONS:
Overall Officials: John JB Allen, PhD, Principal Investigator — University of Arizona

DOCUMENTS (3):
  • Study Protocol (2015-09-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT04023968/Prot_000.pdf
  • Informed Consent Form (2015-09-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT04023968/ICF_001.pdf
  • Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT04023968/SAP_002.pdf